CLINICAL TRIAL: NCT04852081
Title: Analysis of Therapy Sequence in Women With Hormone Receptor-positive, HER2-negative Metastatic Breast Cancer in Russia: A Multicentre Retrospective Observational Real-life Study.
Brief Title: Analysis of Therapy Sequence in Women With HR+, HER2 - mBC in Moscow: A Multicenter Retrospective Observational Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: 01-2021
Record Dates: First submitted 2021-04-11; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer Stage IV
Keywords: HR +, HER2-negative metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; ribociclib; abemaciclib; Letrozole; Anastrozole; Tamoxifen; Fulvestrant; exemestane; Alpelisib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with HR+, HER2- advanced or metastatic breast cancer: patients with HR+, HER2- advanced or metastatic breast cancer
  Interventions: Drug: Palbociclib; Drug: Ribociclib; Drug: Abemaciclib; Drug: Letrozole; Drug: Anastrozole; Drug: Tamoxifen; Drug: Fulvestrant; Drug: Exemestane; Drug: Alpelisib

INTERVENTIONS:
Drug: Palbociclib — Palbociclib is in the form of oral capsules. Palbociclib, capsule, 125 mg taken orally once daily for 21 consecutive days followed by 7 days off treatment to comprise a complete cycle of 28 days. Palbociclib should be taken with food
  Other Names: Ibrance
Drug: Ribociclib — Ribociclib, tablets, 600mg orally (three 200 mg tablets)taken once daily with or without food for 21 consecutive days followed by 7 days off treatment
  Other Names: Kisqali
Drug: Abemaciclib — Abemaciclib in combination with fulvestrant or an aromatase inhibitor: 150 mg twice daily Abemaciclib as monotherapy: 200 mg twice daily. (2.1)
  Other Names: VERZENIO
Drug: Letrozole — Letrozole will be dosed daily at a fixed dose of 2.5 mg/day throughout the study.
Drug: Anastrozole — Anastrozole will be dosed daily at a fixed dose of 1 mg/day throughout the study.
Drug: Tamoxifen — Tamoxifen will be dosed daily at a fixed dose of 20 mg/day throughout the study.
Drug: Fulvestrant — Fulvestrant is in the form of a prefilled syringe containing 5 ml of an injection solution of 250 mg of fulvestrant for intramuscular injection. The recommended dose is once every 28 days, once at a dose of 500 mg, and on the 15th day after the initial injection, a loading dose of fulvestrant 500 mg is added.
  Other Names: Faslodex
Drug: Exemestane — Exemestane will be dosed daily at a fixed dose of 25mg/day throughout the study.
  Other Names: Exemestane will be dosed daily at a fixed dose of 25mg/day throughout the study.
Drug: Alpelisib — Alpelisib will be dosed daily at a fixed dose of 300 mg/day throughout the study.
  Other Names: PIQRAY

SUMMARY:
A assessment of the efficacy of first-/second-line endocrine therapies ± target therapies and chemotherapy in real-life of in patients with hormone receptor-positive (HR+)/HER2-negative metastatic breast cancer has not yet been conducted in Moscow.

Methods: Observational, retrospective study carried out in oncology hospitals in Moscow, in patients with hormone receptor-positive (HR+)/HER2-negative metastatic breast cancer. The descriptive analysis will be conducted for patient characteristics, responses to treatment and treatment outcomes.

This study will provide retrospective chart review of evidence on the use of therapy in routine clinical practice, with a focus in population of Moscow

DETAILED DESCRIPTION:
The combination CDK4/6 inhibitors (CDK4/6i) (Palbociclib, Ribociclib and Abemaciclib) with endocrine therapy (ET, i.e. aro- matase inhibitors (AI) or Fulvestrant) has significantly increased objective response rate (ORR) and progression-free survival (PFS) of first- and second-line treatments in patients with hormone receptor positive, HER2 negative (luminal) mBC. Now this combination is the standard treatment for luminal mBC. Recommendation for endocrine therapy versus chemotherapy as first-line treatment of luminal mBC is endorsed by the main international guidelines such as ASCO and ESO-ESMO guidelines. Endocrine therapy should be used as initial treatment except in cases of immediately life-threatening disease, tumors refractory to endocrine therapy, visceral crisis, or rapid progressive disease that mandate a high response rate treatment. The aim of this study is to provide real-life treatment patterns data for luminal MBC with a focus in population of Moscow

ELIGIBILITY:
Inclusion Criteria:

* Patient has a histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer based on the most recently analyzed tissue sample and all tested by local laboratory. ER should be more than 10% ER positive or Allred ≥5 by local laboratory testing.
* Patient has HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing and based on the most recently analyzed tissue sample.
* Patient has inoperable locally advanced or metastatic breast cancer
* Patient has adequate bone marrow and organ function
* Patient must be physically well enough that they are capable of treatment

Exclusion Criteria:

* Patient has severe acute or chronic medical or psychiatric condition, including recent or active suicidal ideation or behavior, or laboratory abnormality that may interfere with the interpretation of study results
* no clinical and anamnestic information or information about safety or information about effectiveness treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with histologically or cytologically confirmed luminal (HR positive/HER2 negative) inoperable locally advanced or metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
To describe treatment sequences of all lines of therapy received by HER2 + mBC patients in Moscow | 12 months
  The proportion of each type of treatment received for all lines of therapy in the metastatic setting will be determined.

SECONDARY OUTCOMES:
Proportion of patients among study population who have with symptomatic visceral metastasis | 12 months
  Proportion of patients among study population who have with symptomatic visceral metastasis
Proportion of patients among study population who have treatment-emergent Adverse Events | 12 months
  Proportion of patients among study population who have treatment-emergent Adverse Events
Proportion of premenopausal women among study population | 12 months
  Proportion of premenopausal women among study population
percentage of obtaining tumor specimens and reevaluating targeted markers in breast cancer patients who relapsed after curative treatment | 12 months
  percentage of obtaining tumor specimens and reevaluating targeted markers in breast cancer patients who relapsed after curative treatment
Proportion of patients among study population who have visceral metastasis | 12 months
  Proportion of patients among study population who have visceral metastasis
Evaluation of the outcome per treatment line | 12 months
  To evaluate the outcome of patients per treatment line (objective response, progression free survival, time to disease progression per line of therapy), overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Sergei Tjulandin, Principal Investigator — N.N. Blokhin National Medical Research Center of Oncology
Locations (1):
- N.N. Blokhin National Medical Research Center of Oncology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No